CLINICAL TRIAL: NCT01840319
Title: Retrospective Observational Study Of Patients Previously Treated With Tigecycline In ICU And Included In The Previous French Prospective Observational Study
Brief Title: Retrospective Transverse Observational Study Of Previous Study (Initial Protocol, B1811030)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: NRB1810005
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2013-10

CONDITIONS: Survival Status at Day 30 After the Last Intake

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients previously included in the initial protocol WYETH 3074A1-4448 / B1811030. (To collect only status survival data 30 days after the last dose of treatment)

SUMMARY:
The goal of this retrospective observational study is to collect only status survival data 30 days after the last dose of treatment of patients included in the initial protocol WYETH 3074A1-4448 / B1811030. The purpose is to estimate the survival status, 30 days after the last intake of tigecycline to patients hospitalized in ICU and treated by tigecycline.

ELIGIBILITY:
Inclusion Criteria:

* All patients included in the previous study WYETH 3074A1-4448 then Pfizer B1811030 for which mortality status was not known at the closure of this previous study

Exclusion Criteria:

* Patients who has withdrawn their consent for the study WYETH3074A1-4448 then Pfizer B1811030.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients which has already been enrolled in the previous study protocol initial WYETH 3074A1-4448 then Pfizer B1811030
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- France (19):
  - Pfizer Investigational Site, Amiens, France
  - Pfizer Investigational Site, Marseille, France
  - Pfizer Investigational Site, Montpellier, France
  - Pfizer Investigational Site, Paris, France
  - Pfizer Investigational Site, Strasbourg, France
  - Pfizer Investigational Site, Argenteuil
  - Pfizer Investigational Site, Ars-Laquenexy
  - Pfizer Investigational Site, Besançon
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, La Tronche
  - Pfizer Investigational Site, Le Chesnay
  - Pfizer Investigational Site, Le Kremlin-Bicêtre
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Rouen
  - Pfizer Investigational Site, Saint-Etienne
  - Pfizer Investigational Site, Toulouse

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=NRB1810005&StudyName=Retrospective%20Transverse%20Observational%20Study%20Of%20Previous%20Study%20%28Initial%20Protocol%2C%20B1811030%29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed the initial study 3074A1-4448 (B1811030) (NCT00799591) and whose death were not reported at the end of initial study were eligible to participate in the study.
Pre-assignment Details: Out of 156 participants who were enrolled in initial study 3074A1-4448 (B1811030) (NCT00799591), 138 participants did not have dates of death, hence, survival data was retrospectively collected for these participants in this study. All data were then combined with the existing survival data for an updated survival analysis.
Groups:
- Tigecycline: Participants who had received tigecycline, alone or in combination in the initial study, for the treatment of a bacterial infection, were retrospectively observed for survival up to 30 days after last dose of tigecycline.
Period: Overall Study
Arm/Group | Tigecycline
Started | 156
Completed | 156
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants of the initial study 3074A1-4448 (B1811030) (NCT00799591).
Arm/Group | Tigecycline
Number analyzed (Participants) | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Survival at 30 Days After Last Dose of Tigecycline
Description: Survival analysis was calculated using Kaplan-Meier Method. The survival status of participants from the initial study database were collected for survival analysis, if participants did not have the data in the database, the participating clinician requested the vital status information from the center for epidemiology and population health research (CESP). The deceased participants' data were collected and the informed consent form was sent to surviving participants. The existing and the collected survival data were then merged and updated. A survival analysis was performed including a variable treatment period plus 30 follow-up days. The maximum treatment duration observed in the initial study was 78 days. Percentage of participants who were alive at 30 days after last dose (corresponding to Day 108 after first dose of tigecycline) of tigecycline were reported.
Time Frame: 30 days after last dose of Tigecycline (Day 108)
Population: Intent-to-treat (ITT) population included all participants of the initial study 3074A1-4448 (B1811030) (NCT00799591).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tigecycline
Number analyzed (Participants) | 156
percentage of participants | 80.60 [73.04 to 86.24]

ADVERSE EVENTS:
Description: Due to retrospective nature of the study, adverse events data was not collected.
Arm/Group | Tigecycline
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
As this was an observational study therefore, no randomization and control groups were included. This limitation did not allow the comparison of tigecycline treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.